CLINICAL TRIAL: NCT07293793
Title: Pregnancy-Safe Skin Care Guidelines: Expert Consensus Recommendations
Status: Enrolling by invitation | Type: Observational
Sponsor: Venus Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pregnancy-Safe Skin Care-Venus
Record Dates: First submitted 2025-12-06; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy; Skin Care; Dermocosmetics
Keywords: Consensus; Recommendations; Skin Care; Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: A cohort of dermatology and aesthetic medicine experts from the MENA region participating in a Modified Delphi process to develop consensus recommendations on Skin Care dermo cosmetics in Pregnancy

SUMMARY:
This research presents a comprehensive consensus on pregnancy skin care, synthesizing expert recommendations to ensure maternal skin health while prioritizing fetal safety. It outlines safe and effective skin care practices tailored to the physiological and hormonal changes during pregnancy. Key guidelines emphasize the use of gentle cleansing, adequate hydration, mineral-based sun protection, and the selection of dermatologically safe ingredients such as vitamin C, hyaluronic acid, niacinamide, and azelaic acid. The consensus highlights the avoidance of potentially harmful substances including retinoids, high-dose salicylic acid, and certain chemical sunscreens. Additionally, the research provides clinical guidance on managing common pregnancy-related skin conditions and cautions against aggressive cosmetic procedures. The outcomes serve as a critical resource for dermatologists and healthcare providers to optimize skin care regimens during pregnancy, balancing efficacy with safety for both mother and child.

DETAILED DESCRIPTION:
Background and Rationale

Pregnancy is associated with profound hormonal, immunological, and metabolic changes that directly affect the skin. These changes can manifest as physiologic alterations (e.g., hyperpigmentation, striae), exacerbation of pre-existing dermatologic diseases, or pregnancy-specific dermatoses. Safe and effective skin care during pregnancy is critical, as many commonly used dermatologic ingredients cross the placental barrier, lack human safety data, or pose teratogenic risks.

Despite the high prevalence of dermatologic concerns in pregnancy, current clinical guidance remains fragmented, variable across regions, and often based on expert opinion rather than standardized consensus. To address this gap, we employed a structured Delphi expert consensus process to develop evidence-informed, practical, and regionally adaptable guidelines for pregnancy-safe skin care.

Methods: Delphi Consensus Process

A structured three-round Delphi methodology was used to achieve consensus among a multidisciplinary panel of dermatologists, obstetricians, and pharmacology experts.

2.1. Panel Composition

N = 25 experts

Representatives from dermatology, maternal-fetal medicine, and clinical pharmacology

Minimum of 5 years of clinical experience

Geographic representation from MENA, Europe, and Asia

Steps in the Delphi Process Round 1: Exploration

Experts provided open-ended responses on:

Essential principles of pregnancy-safe skin care

Ingredient safety classifications

Preferred management of common dermatologic conditions

Cultural and regional care considerations

A qualitative analysis was performed to derive core themes.

Round 2: Structured Statements

75 draft statements were generated and rated using a 9-point Likert scale

1-3: Disagree

4-6: Uncertain

7-9: Agree

Consensus defined as ≥ 75% of experts rating 7-9.

Round 3: Refinement and Final Voting

Statements near consensus were revised for clarity.

Final voting achieved consensus on statements, forming the basis of the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified dermatologist or plastic surgeon OR physician practicing aesthetic medicine.

  * Minimum of 5 years of clinical experience.
  * Practicing within Egypt or the Middle East and North Africa (MENA) region.
  * Willingness to participate in Delphi rounds and provide expert ratings.
  * Ability to read and respond to surveys in English.

Exclusion Criteria:

Inability or unwillingness to complete Delphi rounds.

* Lack of clinical experience with Pregnant ladies.
* Industry representatives without direct clinical practice.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: e study population consisted of a multidisciplinary panel of experts selected to represent diverse clinical, academic, and regional perspectives relevant to dermatologic care during pregnancy to ensure comprehensive evaluation of skin care ingredient safety, therapeutic practices, and procedure-related considerations for pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Achievement of Expert Consensus on Pregnancy-Safe Skin Care Recommendations | 6-12 weeks
  The primary outcome of this Delphi study was to establish consensus-based, evidence-aligned recommendations for safe skin care practices, cosmetic ingredients, and dermatologic treatments during pregnancy. Consensus was defined a priori as:
  ≥75% of experts scoring a statement 7-9 on a 9-point Likert scale (agreement),
  with a median score ≥7.
  This outcome reflects the degree to which experts converged on the safety categories, usage guidelines, and clinical management strategies for skin care in pregnant patients.

SECONDARY OUTCOMES:
Classification of Dermatologic Ingredients and Procedures According to Safety Profile | 6-12 weeks
  A key secondary outcome was the categorization of commonly used dermatologic and cosmetic components into:
  Safe
  Use with Caution (insufficient or limited evidence)
  Avoid (potential teratogenic risk or high systemic absorption)
  This includes topical ingredients, professional procedures, and over-the-counter skin care actives.

CONTACTS AND LOCATIONS:
Locations (1):
- Venus Research Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Delphi studies do not collect patient data, medical records, biological samples, or identifiable clinical information. Experts only give opinions, not "IPD." Their responses are anonymized, and sharing identifiable expert-level responses is not required and often discouraged